CLINICAL TRIAL: NCT02213042
Title: An Open-Label, Phase II, Study to Evaluate Biomarkers Associated With Response to Subsequent Therapies in Subjects With HER2-Positive Metastatic Breast Cancer Receiving Treatment With Trastuzumab in Combination With Lapatinib or Chemotherapy (EGF117165)
Brief Title: Evaluation of Biomarkers Associated With Response to Subsequent Therapies in Subjects With HER2-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary analysis was completed in 2018 and continued minimal data collection from the one participant active in the study was not expected to add meaningful knowledge to the understanding of lapatinib
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117165; 2014-001220-30 (EudraCT Number); CLAP016A2206 (Other: Novartis)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Neoplasms, Breast
Keywords: CLAP016A2206; biomarker; Lapatinib; Prosigna; ErbB2; PAM50; HER2; HER2-overexpressing metastatic breast cancer; HER2-enriched; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Aromatase Inhibitors

STUDY DESIGN:
Intervention Model Description: Participants were randomized to Arms A and B but randomized to Arm C.
Masking Description: This was a two-cohort, three-arm, open-label Phase II study to evaluate the changes in the expression of biomarkers between pre-treatment and progression biopsy in subjects with Human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer. Subjects were allocated to 1 of 2 cohorts depending on the molecular subtype of their biopsy.
  Cohort 1 HER2 -enriched included HER2-positive subjects with a HER2-Enriched molecular subtype, and were randomized in a 1:1 ratio to receive either trastuzumab in combination with lapatinib (Arm A) or trastuzumab in combination with chemotherapy (Arm B).
  Cohort 2 non-HER2-enriched, included HER2-positive subjects with luminal A, luminal B, and basal-like molecular subtypes and were to receive trastuzumab in combination with lapatinib (Arm C). Subjects with hormone receptor (ER and/or PgR)-positive MBC in this arm were required to be treated with an AI of the Investigator's choice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lapatinib 1000mg + Trastuzumab in HER2 Enriched (Active Comparator): In subjects with HER2-overexpressing MBC with a molecular subtype of HER2 Enriched, Lapatinib 1000mg once daily orally along with Trastuzumab (loading dose of 8 milligram/ kilogram (mg/kg) followed by the maintenance dose of 6 mg/kg Intravenous (IV) Every 3 weeks (q3weekly)) or Lapatinib 1000 milligram (mg) once daily orally along with Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly. For subjects who were hormone receptor positive, an aromatase inhibitor of the investigator's choice was required.
  Interventions: Drug: Lapatinib; Biological: Trastuzumab; Drug: Aromatase Inhibitors (AIs)
- Trastuzumab in HER2 Enriched (Active Comparator): In subjects with HER2-overexpressing MBC with a molecular subtype of HER2 Enriched, Trastuzumab (loading dose of 8 mg/kg followed by the maintenance dose of 6 mg/kg IV q3weekly) along with chemotherapy of the investigator's choice or Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly along with chemotherapy of the investigators choice. Subjects randomized to this arm and hormone receptor positive received an aromatase inhibitor at the discretion of the investigator.
  Interventions: Biological: Trastuzumab; Drug: Aromatase Inhibitors (AIs)
- Lapatinib 1000mg + Trastuzumab in Non- HER2 Enriched (Active Comparator): In subjects with HER2-overexpressing MBC with a molecular subtype of Non- HER2 Enriched (luminal A, luminal B or Basal type), Lapatinib 1000mg once daily orally along with Trastuzumab (loading dose of 8 milligram/ kilogram (mg/kg) followed by the maintenance dose of 6 mg/kg Intravenous (IV) Every 3 weeks (q3weekly)) or Lapatinib 1000 milligram (mg) once daily orally along with Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly. For subjects who were hormone receptor positive, an aromatase inhibitor of the investigator's choice was required.
  Interventions: Drug: Lapatinib; Biological: Trastuzumab; Drug: Aromatase Inhibitors (AIs)

INTERVENTIONS:
Drug: Lapatinib — Lapatinib is available as 250-mg orange tablets. Subjects randomized to the Lapatinib plus Trastuzumab arm received 1000 mg per day of Lapatinib, so wre instructed to take 4 x 250 mg tablets per day. Lapatinib was to be taken either 1 hour (or more) before a meal or 1 hour (or more) after a meal
  Arms: Lapatinib 1000mg + Trastuzumab in HER2 Enriched; Lapatinib 1000mg + Trastuzumab in Non- HER2 Enriched
Biological: Trastuzumab — Trastuzumab is a sterile, white to pale yellow, preservative-free lyophilized powder for IV administration. Trastuzumab was administered on Day 1 of the start of Lapatinib or in conjunction with the first cycle of chemotherapy, as an 8 mg/kg loading dose. Subsequently, Trastuzumab was administered q3weekly as a 6 mg/kg maintenance dose. At the discretion of the investigator, weekly Trastuzumab could be given in either of the three treatment arms (loading dose 4mg/kg followed by weekly administration of 2mg/kg).
Drug: Aromatase Inhibitors (AIs) — Subjects who were hormone receptor-positive were required to receive an aromatase inhibitor as combination treatment; however the choice of the aromatase inhibitor selected for each patient was determined by the patients' investigator. The AIs the Investigator could choose from were anastrozole, exemestane, and letrozole and dosing was per product information.

SUMMARY:
This was a multicenter, open-label, Phase II study in subjects with Human epidermal growth factor receptor (HER2)-positive metastatic breast cancer who received at least 2 prior lines of anti-HER2-targeted therapies of which at least one included a Trastuzumab-containing regimen. This study was a post-approval commitment with regulatory authorities. It was designed to evaluate whether treatment with Dual blockade promoted changes to biomarkers associated with immunomodulation.

DETAILED DESCRIPTION:
This study was designed to address the post-authorization measures as agreed with the Committee for Medicinal Products for Human Use (CHMP). Recruitment of subjects into this study was challenging, and following agreement with the European Medicines Agency (EMA) enrollment into this study was halted after the enrollment of 42 of the 225 planned subjects.

The primary endpoint of the study evaluated changes in expression of biomarkers associated with immunomodulation between a pre-treatment biopsy and the disease progression biopsy. Secondary efficacy endpoints included overall response rate, clinical benefit rate and progression-free survival (PFS), as well as safety/tolerability. All subjects received study treatment until disease progression, death, unacceptable toxicity, or subject withdrawal. In case of disease progression during the treatment period, the subject was followed-up for 30 days for safety evaluation. In case of study treatment discontinuation for any reasons other than disease progression, the subject was followed-up for safety and efficacy assessments until disease progression, new anticancer therapy, death, withdrawal of consent or end of study, whichever came first.

This study supported a better understanding of the rapidly accumulating evidence for the importance of the immune microenvironment in HER2-positive breast cancer and the observed immunomodulation in the neoadjuvant setting could be confirmed in the advanced setting and supported the putative mechanism of action of HER2 dual blockade and its potential function on the tumor microenvironment. No formal comparisons between treatment arms were undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Female >=18 years
* Histologically or cytologically confirmed invasive breast cancer with distant metastasis
* Subjects must have at least one measurable lesion per RECIST 1.1
* Note: Biopsied lesions should not be used as target lesions.
* Documentation of HER2 overexpression or gene amplification, in the invasive component of either the primary tumor or metastatic disease site as defined as: 3+ by Immunohistochemistry (IHC) and/or
* HER2/neu gene amplification by fluorescence, chromogenic, or silver in situ hybridization [FISH, CISH or SISH;>=6 HER2/neu gene copies per nucleus or a FISH, CISH, or SISH test ratio (HER2 gene copies to chromosome 17 signals) of >=2.0 OR HER2/chromosome 17 ratio <=2.0 with average HER2 copy number >=6 signals/cell nucleus]
* Centrally determined HER2-positive, hormone receptor status, breast molecular subtype by Prediction Analysis of Microarray 50 (PAM50) on the pre-treatment biopsy of metastatic lesion obtained during screening
* Note: Biopsied lesions should not be used as target lesions.
* Progression on at least 2 lines of anti-HER2-targeted therapies for metastatic breast cancer (MBC)
* Documented radiological disease progression during the most recent treatment regimen for metastatic disease
* Most recent treatment regimen for metastatic disease must include Trastuzumab and chemotherapy.
* Note: Trastuzumab emtansine (T-DM1) is considered acceptable as prior Trastuzumab/chemotherapy regimen
* Agreement to provide 2 tumor biopsies
* Prior treatment with pertuzumab, Lapatinib, and/or Trastuzumab emtansine is allowed; however, the last treatment for MBC must not include Trastuzumab in combination with pertuzumab.
* Subjects with radiographically stable Central nervous system (CNS) metastases, defined as radiographically stable on the previous 2 brain imaging scans, asymptomatic, and off systemic steroids and anticonvulsants for at least 1 month are eligible; treatment with prophylactic anticonvulsants is permitted unless listed under Prohibited Medications
* Discontinuation of all prior chemotherapy, immunotherapy, or biological therapy at least 3 weeks prior to the first dose of investigational product is required.
* Note: Discontinuation of Trastuzumab is not necessary.
* All treatment related toxicities, except alopecia, must have recovered to Grade 1 or better (Common Terminology Criteria for Adverse Events (CTCAE); version 4.0) prior to administration of the first dose of study treatment.
* Baseline Left ventricular ejection fraction (LVEF) >=50% as measured by Echocardiogram (ECHO) or Multigated acquisition (MUGA) and above the testing institution's lower limit of normal
* QT interval corrected (QTc) <450 millisecond (msec) or QTc <480 msec for patients with bundle branch block.
* The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB)
* Fridericia's formula (QTcF), or another method, machine or manual overread.
* For subject eligibility and withdrawal, QT correction formula QTcB will be used.
* For purposes of this data analysis, Bazett's formula will be used as the primary method of calculating the corrected QT interval. The QTc should be based on either a single Electrocardiogram (ECG) or an average of 3 sequential ECGs obtained within 24 hours of each other.
* The QTc should be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment and agree to use effective contraception, during the study and for 30 days following the last dose of study treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Completion of screening and baseline assessments
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* At least 4 weeks must have elapsed since the last surgery and 2 weeks must have elapsed since radiotherapy
* Adequate baseline organ function as defined below
* Screening laboratory values should be used to confirm subject eligibility. Laboratory results may be retested if necessary to confirm eligibility.
* Hematologic(These values must be independent of growth factor support and stable for at least one week post transfusion)
* Absolute neutrophil count >=1.5 x 10^9/litre (L)
* Hemoglobin >=9.0 grams/decilitre(g/dL) (after transfusion if needed)
* Platelets>=100 x 10^9/L
* Hepatic
* Albumin >=2.5 g/dL
* Serum bilirubin <=1.25 x upper limit of normal (ULN)( These values must be independent of growth factor support and stable for at least one week post transfusion)
* Alanine aminotransferase; and, Aspartate aminotransferase AST and ALT<=2.5 x ULN
* Renal
* Calculate creatinine clearance >=40 millilitre/ minute (mL/min) (With the exception of those subjects who have Gilbert's syndrome; the bilirubin in these subjects should be at their baseline)

Exclusion Criteria:

* Lactating female
* Note: Women with potential to have children must be willing to practice acceptable methods of birth control during the study
* Bone-only disease and/or disease that cannot be biopsied.
* Unstable CNS metastases or leptomeningeal carcinomatosis not considered radiographically stable
* Note: Subjects with radiographically stable CNS metastases are defined as radiographically stable on the previous 2 brain imaging studies, asymptomatic, and off systemic steroids and anticonvulsants for at least 1 month; treatment with prophylactic anticonvulsants is permitted unless listed under prohibited medications
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions including concurrent disease that could interfere with subject's safety, obtaining informed consent, or compliance with the study procedures.
* Serious cardiac illness or medical condition including but not confined to: Uncontrolled arrhythmias (e.g. ventricular tachycardia, high-grade atrioventricular (AV)-block, supraventricular arrhythmias which are not adequately rate-controlled);
* Angina pectoris requiring antianginal medication
* History of congestive heart failure or systolic dysfunction (LVEF <50%)
* Documented myocardial infarction <6 months from study entry
* Evidence of transmural infarction on ECG
* Poorly controlled hypertension (e.g. systolic >160milimiter (mm) Mercury (Hg) or diastolic >100mm Hg)
* Clinically significant valvular heart disease
* Current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment)
* Any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels as well as subjects with ulcerative colitis are also excluded
* Any prohibited medication
* Prior treatment with Trastuzumab in combination with Lapatinib or prior treatment with an irreversible inhibitor of the intracellular domain of the HER2 receptor such as neratinib
* Last treatment for metastatic disease including Trastuzumab in combination with pertuzumab
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study drugs or their excipients that, in the opinion of the investigator or medical monitor, contraindicates participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (3):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Houston, Texas
- Argentina (8):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Viedma, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Rioja
  - Novartis Investigative Site, San Miguel de Tucumán
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Brazil (7):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São José do Rio Preto
- Hong Kong (2):
  - Novartis Investigative Site, Pok Fu Lam
  - Novartis Investigative Site, Pokfulam
- Novartis Investigative Site, Milan, Lombardy, Italy
- Novartis Investigative Site, México, Mexico
- Peru (2):
  - Novartis Investigative Site, Arequipa
  - Novartis Investigative Site, Lima
- Philippines (2):
  - Novartis Investigative Site, Cebu
  - Novartis Investigative Site, Manila
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Volzhskiy
- Spain (6):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Phitsanulok

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 225 subjects were planned and 42 subjects were enrolled in this study
Pre-assignment Details: This study was designed to address the post-authorization measures as agreed with the Committee for Medicinal Products for Human Use (CHMP). Recruitment of subjects into this study was challenging, and following agreement with the European Medicines Agency (EMA) enrollment into this study was halted after the enrollment of 42 of the 225 planned subjects.
Groups:
- LAP+TRAS±AI (HER2-Enriched) - Arm A: Lapatinib 1000mg + Trastuzumab in HER2 Enriched In subjects with HER2-overexpressing MBC with a molecular subtype of HER2 Enriched, Lapatinib 1000mg once daily orally along with Trastuzumab (loading dose of 8 milligram/ kilogram (mg/kg) followed by the maintenance dose of 6 mg/kg Intravenous (IV) Every 3 weeks (q3weekly)) or Lapatinib 1000 milligram (mg) once daily orally along with Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly. For subjects who were hormone receptor positive, an aromatase inhibitor of the investigator's choice was required.
- TRAS+CHEM±AI (HER2-Enriched) - Arm B: Trastuzumab in HER2 Enriched: In subjects with HER2-overexpressing MBC with a molecular subtype of HER2 Enriched, Trastuzumab (loading dose of 8 mg/kg followed by the maintenance dose of 6 mg/kg IV q3weekly) along with chemotherapy of the investigator's choice or Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly along with chemotherapy of the investigators choice. Subjects randomized to this arm and hormone receptor positive received an aromatase inhibitor at the discretion of the investigator.
- Non-HER2- Enriched - Arm C: Lapatinib 1000mg + Trastuzumab in Non- HER2 Enriched: In subjects with HER2-overexpressing MBC with a molecular subtype of Non- HER2 Enriched (luminal A, luminal B or Basal type), Lapatinib 1000mg once daily orally along with Trastuzumab (loading dose of 8 milligram/ kilogram (mg/kg) followed by the maintenance dose of 6 mg/kg Intravenous (IV) Every 3 weeks (q3weekly)) or Lapatinib 1000 milligram (mg) once daily orally along with Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly. For subjects who were hormone receptor positive, an aromatase inhibitor of the investigator's choice was required.
Period: Overall Study
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Started | 17 | 15 | 10
Total Deaths | 11 | 9 | 6
Completed | 0 | 0 | 0
Not Completed | 17 | 15 | 10
Not completed — Disease progression (incl. death due to disease progression) | 14 | 13 | 8
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Consisted of all subjects who were randomized to study Arm A or Arm B or assigned to study Arm C, irrespective of whether they actually received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C | Total
Number analyzed (Participants) | 17 | 15 | 10 | 42
Age, Customized [Number; unit: Participants]
  < 65 years | 14 | 15 | 6 | 35
  >= 65 years | 3 | 0 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 10 | 42
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 14 | 11 | 10 | 35
  African American | 1 | 2 | 0 | 3
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Expression Profile of Genes and/or Proteins for Arm A (LAP+TRAS±AI (HER2-Enriched)) From Screening to Approx. 3.5 Years
Description: Evaluate changes in biomarkers associated with immunomodulation between pre-treatment biopsy and disease progression biopsy within each arm. Biomarker analysis was performed using an mRNA gene expression panel derived from Nanostring platform in a total of 20 subjects who received the study treatment as per the study design and with baseline tumor biopsies available.
  For the selected biomarkers associated with immunomodulation, the median fold changes of gene expression level and 95% confidence interval are presented. The fold change was calculated as the ratio of the expression level of a biomarker at disease progression over the baseline.
Time Frame: At screening and at disease progression, assessed up to approx. 3.5 years
Population: Evaluable Set: Included all subjects in Arm A who received the study treatment and had both baseline and progression tumor biopsies available, with evaluable data for at least 1 biomarker.
Measure: Median (95% Confidence Interval); unit: Ratio of gene expression level
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A
Number analyzed (Participants) | 7
Ratio of gene expression level
  Membrane spanning 4-domains A1: number analyzed (Participants) | 5
  Membrane spanning 4-domains A1 | 0.25 [0.078 to 0.589]
  POU class 2 associating factor 1: number analyzed (Participants) | 5
  POU class 2 associating factor 1 | 0.32 [0.183 to 0.543]
  CD19+: number analyzed (Participants) | 5
  CD19+ | 0.35 [0.106 to 0.904]
  Interleukin 6: number analyzed (Participants) | 5
  Interleukin 6 | 0.36 [0.033 to 0.832]
  G antigen 1: number analyzed (Participants) | 5
  G antigen 1 | 0.43 [0.030 to 0.901]
  ubiquitin specific peptidase 9, Y-linked: number analyzed (Participants) | 5
  ubiquitin specific peptidase 9, Y-linked | 0.50 [0.321 to 0.770]
  Thy-1 cell surface antigen: number analyzed (Participants) | 5
  Thy-1 cell surface antigen | 0.50 [0.113 to 0.902]
  Chemerin chemokine-like receptor 1: number analyzed (Participants) | 5
  Chemerin chemokine-like receptor 1 | 0.51 [0.345 to 0.862]
  Major histocompatibility complex, class II, DR beta 4: number analyzed (Participants) | 5
  Major histocompatibility complex, class II, DR beta 4 | 0.51 [0.320 to 0.984]
  Collectin subfamily member 12: number analyzed (Participants) | 5
  Collectin subfamily member 12 | 0.51 [0.151 to 0.794]
  Complement C3b/C4b receptor 1 (Knops blood group): number analyzed (Participants) | 5
  Complement C3b/C4b receptor 1 (Knops blood group) | 0.51 [0.227 to 0.901]
  CD33 molecule: number analyzed (Participants) | 5
  CD33 molecule | 0.56 [0.458 to 0.826]
  B-cell linker: number analyzed (Participants) | 5
  B-cell linker | 0.56 [0.326 to 0.874]
  Interleukin 12A: number analyzed (Participants) | 5
  Interleukin 12A | 0.57 [0.228 to 0.892]
  CD163+: number analyzed (Participants) | 5
  CD163+ | 0.57 [0.417 to 0.911]
  C-C motif chemokine ligand 8: number analyzed (Participants) | 5
  C-C motif chemokine ligand 8 | 0.58 [0.138 to 0.954]
  Chemokine (C-C motif) receptor 1: number analyzed (Participants) | 5
  Chemokine (C-C motif) receptor 1 | 0.59 [0.501 to 0.792]
  POU class 2 homeobox 2: number analyzed (Participants) | 5
  POU class 2 homeobox 2 | 0.60 [0.440 to 0.944]
  Cyclin dependent kinase inhibitor 1A: number analyzed (Participants) | 5
  Cyclin dependent kinase inhibitor 1A | 0.62 [0.453 to 0.873]
  CD27 molecule: number analyzed (Participants) | 5
  CD27 molecule | 0.62 [0.357 to 0.886]
  Lymphocyte antigen 86: number analyzed (Participants) | 5
  Lymphocyte antigen 86 | 0.63 [0.383 to 0.906]
  TNF superfamily member 8: number analyzed (Participants) | 5
  TNF superfamily member 8 | 0.64 [0.476 to 0.879]
  CD34+: number analyzed (Participants) | 5
  CD34+ | 0.67 [0.558 to 0.863]
  Integrin subunit alpha 6: number analyzed (Participants) | 5
  Integrin subunit alpha 6 | 0.68 [0.470 to 0.827]
  C-type lectin domain containing 7A: number analyzed (Participants) | 5
  C-type lectin domain containing 7A | 0.69 [0.326 to 0.944]
  CD180 molecule: number analyzed (Participants) | 5
  CD180 molecule | 0.70 [0.347 to 0.869]
  Integrin subunit alpha M: number analyzed (Participants) | 5
  Integrin subunit alpha M | 0.72 [0.411 to 0.957]
  Toll like receptor 6: number analyzed (Participants) | 5
  Toll like receptor 6 | 0.72 [0.511 to 0.836]
  Autophagy related 10: number analyzed (Participants) | 5
  Autophagy related 10 | 0.73 [0.662 to 0.864]
  C-C motif chemokine ligand 3 like 1: number analyzed (Participants) | 5
  C-C motif chemokine ligand 3 like 1 | 0.74 [0.499 to 0.996]
  Bone marrow stromal cell antigen 1: number analyzed (Participants) | 5
  Bone marrow stromal cell antigen 1 | 0.75 [0.345 to 0.922]
  CD22+: number analyzed (Participants) | 5
  CD22+ | 0.76 [0.629 to 0.936]
  CD37 molecule: number analyzed (Participants) | 5
  CD37 molecule | 0.76 [0.553 to 0.884]
  NEG_A: number analyzed (Participants) | 5
  NEG_A | 0.77 [0.674 to 0.949]
  Sperm auto antigenic protein 17: number analyzed (Participants) | 5
  Sperm auto antigenic protein 17 | 0.79 [0.697 to 0.968]
  CD200 molecule: number analyzed (Participants) | 5
  CD200 molecule | 0.79 [0.598 to 0.945]
  TNF receptor associated factor 3: number analyzed (Participants) | 5
  TNF receptor associated factor 3 | 0.82 [0.718 to 0.962]
  Interferon alpha and beta receptor subunit 1: number analyzed (Participants) | 5
  Interferon alpha and beta receptor subunit 1 | 1.10 [1.036 to 1.124]
  TNF receptor associated factor 6: number analyzed (Participants) | 5
  TNF receptor associated factor 6 | 1.21 [1.016 to 1.332]

2. Primary Outcome: Fold Change in Expression Profile of Genes and /or Proteins for Arm B (TRAS+CHEM±AI (HER2-Enriched)) From Screening to Approx. 3.5 Years
Description: as for outcome 1
Time Frame: At screening and at disease progression, assessed up to approx. 3.5 years
Population: Evaluable Set: Included all subjects in Arm B who received the study treatment and had both baseline and progression tumor biopsies available, with evaluable data for at least 1 biomarker.
Measure: Median (95% Confidence Interval); unit: Ratio of gene expression level
Arm/Group | TRAS+CHEM±AI (HER2-Enriched) - Arm B
Number analyzed (Participants) | 6
Ratio of gene expression level
  C-type lectin domain containing 5A: number analyzed (Participants) | 5
  C-type lectin domain containing 5A | 0.16 [0.020 to 0.440]
  Interferon induced transmembrane protein 1: number analyzed (Participants) | 5
  Interferon induced transmembrane protein 1 | 0.25 [0.183 to 0.421]
  Fibronectin 1: number analyzed (Participants) | 5
  Fibronectin 1 | 0.27 [0.077 to 0.393]
  C-C motif chemokine ligand 7: number analyzed (Participants) | 5
  C-C motif chemokine ligand 7 | 0.27 [-0.064 to 0.888]
  Triggering receptor expressed on myeloid cells 1: number analyzed (Participants) | 5
  Triggering receptor expressed on myeloid cells 1 | 0.27 [-0.018 to 0.959]
  Plasminogen activator, urokinase: number analyzed (Participants) | 5
  Plasminogen activator, urokinase | 0.27 [0.112 to 0.545]
  Interleukin 22 receptor subunit alpha 2: number analyzed (Participants) | 5
  Interleukin 22 receptor subunit alpha 2 | 0.28 [0.192 to 0.425]
  C-C motif chemokine ligand 8: number analyzed (Participants) | 5
  C-C motif chemokine ligand 8 | 0.28 [0.044 to 0.699]
  Tumor necrosis factor (ligand) superfamily member 4 gene: number analyzed (Participants) | 5
  Tumor necrosis factor (ligand) superfamily member 4 gene | 0.31 [0.147 to 0.651]
  Major histocompatibility complex, Class I-related: number analyzed (Participants) | 5
  Major histocompatibility complex, Class I-related | 0.32 [0.139 to 0.832]
  Cathepsin L: number analyzed (Participants) | 5
  Cathepsin L | 0.32 [0.066 to 0.820]
  SPP-1 (Osteopontin): number analyzed (Participants) | 5
  SPP-1 (Osteopontin) | 0.33 [0.076 to 0.501]
  Thy-1 cell surface antigen: number analyzed (Participants) | 5
  Thy-1 cell surface antigen | 0.34 [0.157 to 0.648]
  Transforming growth factor beta 2: number analyzed (Participants) | 5
  Transforming growth factor beta 2 | 0.35 [0.120 to 0.504]
  Hepatitis A virus cellular receptor 2: number analyzed (Participants) | 5
  Hepatitis A virus cellular receptor 2 | 0.36 [0.138 to 0.614]
  Bone marrow stromal cell antigen 1: number analyzed (Participants) | 5
  Bone marrow stromal cell antigen 1 | 0.37 [0.133 to 0.864]
  C-type lectin domain containing 7A: number analyzed (Participants) | 5
  C-type lectin domain containing 7A | 0.37 [0.166 to 0.570]
  C-X-C motif chemokine ligand 5: number analyzed (Participants) | 5
  C-X-C motif chemokine ligand 5 | 0.38 [0.040 to 0.943]
  Collagen type III alpha 1 chain: number analyzed (Participants) | 5
  Collagen type III alpha 1 chain | 0.40 [0.130 to 0.685]
  Complement C1s: number analyzed (Participants) | 5
  Complement C1s | 0.41 [0.088 to 0.717]
  IFIT1 gene: number analyzed (Participants) | 5
  IFIT1 gene | 0.41 [0.148 to 0.921]
  Major histocompatibility complex, class I, G: number analyzed (Participants) | 5
  Major histocompatibility complex, class I, G | 0.41 [0.147 to 0.698]
  Tumour necrosis factor gene: number analyzed (Participants) | 5
  Tumour necrosis factor gene | 0.42 [0.108 to 0.945]
  Integrin subunit beta 1: number analyzed (Participants) | 5
  Integrin subunit beta 1 | 0.43 [0.231 to 0.864]
  Pro-melanin concentrating hormone: number analyzed (Participants) | 5
  Pro-melanin concentrating hormone | 0.43 [0.081 to 0.972]
  CD86+: number analyzed (Participants) | 5
  CD86+ | 0.44 [0.102 to 0.700]
  FCGR3A SNP rs396991: number analyzed (Participants) | 5
  FCGR3A SNP rs396991 | 0.44 [0.107 to 0.696]
  TNF receptor superfamily member 10c: number analyzed (Participants) | 5
  TNF receptor superfamily member 10c | 0.44 [0.165 to 0.925]
  Integrin subunit alpha M: number analyzed (Participants) | 5
  Integrin subunit alpha M | 0.45 [0.166 to 0.797]
  TNF receptor superfamily member 11b: number analyzed (Participants) | 5
  TNF receptor superfamily member 11b | 0.45 [0.114 to 0.923]
  Platelet derived growth factor C: number analyzed (Participants) | 5
  Platelet derived growth factor C | 0.45 [0.231 to 0.797]
  Mannan binding lectin serine peptidase 1: number analyzed (Participants) | 5
  Mannan binding lectin serine peptidase 1 | 0.46 [0.304 to 0.896]
  Recombination activating 1: number analyzed (Participants) | 5
  Recombination activating 1 | 0.46 [0.394 to 0.597]
  Interleukin 22: number analyzed (Participants) | 5
  Interleukin 22 | 0.47 [0.229 to 0.609]
  Tumor necrosis factor (ligand) superfamily member 13b gene: number analyzed (Participants) | 5
  Tumor necrosis factor (ligand) superfamily member 13b gene | 0.47 [0.179 to 0.697]
  BMI1 proto-oncogene, polycomb ring finger: number analyzed (Participants) | 5
  BMI1 proto-oncogene, polycomb ring finger | 0.47 [0.322 to 0.735]
  CXCL10 gene: number analyzed (Participants) | 5
  CXCL10 gene | 0.48 [0.074 to 0.986]
  Leukocyte immunoglobulin like receptor B1: number analyzed (Participants) | 5
  Leukocyte immunoglobulin like receptor B1 | 0.48 [0.142 to 0.747]
  MX1 gene: number analyzed (Participants) | 5
  MX1 gene | 0.48 [0.155 to 0.781]
  Tumor necrosis factor (ligand) superfamily member 11 gene: number analyzed (Participants) | 5
  Tumor necrosis factor (ligand) superfamily member 11 gene | 0.48 [0.227 to 0.798]
  Cathepsin S: number analyzed (Participants) | 5
  Cathepsin S | 0.49 [0.138 to 0.807]
  Interferon induced transmembrane protein 2: number analyzed (Participants) | 5
  Interferon induced transmembrane protein 2 | 0.49 [0.245 to 0.887]
  LYN proto-oncogene, Src family tyrosine kinase: number analyzed (Participants) | 5
  LYN proto-oncogene, Src family tyrosine kinase | 0.50 [0.360 to 0.685]
  Platelet derived growth factor receptor beta: number analyzed (Participants) | 5
  Platelet derived growth factor receptor beta | 0.50 [0.160 to 0.801]
  OAS3 gene: number analyzed (Participants) | 5
  OAS3 gene | 0.50 [0.284 to 0.899]
  CD58 molecule: number analyzed (Participants) | 5
  CD58 molecule | 0.50 [0.398 to 0.619]
  complement C3a receptor 1: number analyzed (Participants) | 5
  complement C3a receptor 1 | 0.51 [0.147 to 0.949]
  Chemokine (C-C motif) receptor 1: number analyzed (Participants) | 5
  Chemokine (C-C motif) receptor 1 | 0.52 [0.159 to 0.815]
  Interleukin 24 gene: number analyzed (Participants) | 5
  Interleukin 24 gene | 0.52 [0.161 to 0.706]
  Chemokine (C-X-C motif) receptor 2: number analyzed (Participants) | 5
  Chemokine (C-X-C motif) receptor 2 | 0.53 [0.295 to 0.629]
  Strawberry notch homolog 2: number analyzed (Participants) | 5
  Strawberry notch homolog 2 | 1.13 [1.045 to 1.300]
  Zinc finger protein 205: number analyzed (Participants) | 5
  Zinc finger protein 205 | 1.42 [1.144 to 1.815]
  Fas associated via death domain: number analyzed (Participants) | 5
  Fas associated via death domain | 1.58 [1.107 to 2.043]
  CD3e molecule associated protein: number analyzed (Participants) | 5
  CD3e molecule associated protein | 1.67 [1.244 to 2.075]
  Baculoviral IAP repeat containing 5: number analyzed (Participants) | 5
  Baculoviral IAP repeat containing 5 | 1.73 [1.003 to 2.635]
  Interleukin 17 receptor B: number analyzed (Participants) | 5
  Interleukin 17 receptor B | 2.01 [1.151 to 2.975]

3. Primary Outcome: Fold Change in Expression Profile of Genes and /or Proteins for Arm C (Non-HER2- Enriched) From Screening to Approx. 3.5 Years
Description: as for outcome 1
Time Frame: At screening and at disease progression, assessed up to approx. 3.5 years
Population: Evaluable Set: Included all subjects in Arm C who received the study treatment and had both baseline and progression tumor biopsies available, with evaluable data for at least 1 biomarker.
Measure: Median (95% Confidence Interval); unit: Ratio of gene expression level
Arm/Group | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 7
Ratio of gene expression level
  Triggering receptor expressed on myeloid cells 1: number analyzed (Participants) | 5
  Triggering receptor expressed on myeloid cells 1 | 0.50 [0.294 to 0.995]
  Interleukin 1 receptor, type 1 gene: number analyzed (Participants) | 5
  Interleukin 1 receptor, type 1 gene | 1.58 [1.235 to 2.328]
  Complement component 2: number analyzed (Participants) | 5
  Complement component 2 | 2.13 [1.011 to 3.567]
  Coagulation factor XII: number analyzed (Participants) | 5
  Coagulation factor XII | 2.69 [1.062 to 4.229]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization (for Arm A and B) / treatment start date (for Arm C) to the date of the first documented disease progression or death due to any cause, whichever was earlier. If a subject had not progressed or died at the analysis cutoff date, PFS was censored at the time of the last adequate tumor assessment. PFS was summarized using Kaplan-Meier estimates.
Time Frame: From randomization to disease progression or death, up to approx. 5.6 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 17 | 15 | 10
Months | 6.0 [2.10 to 10.60] | 7.2 [2.10 to 14.80] | 6.0 [1.60 to 8.30]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of subjects achieving either a confirmed complete response (CR) or partial response (PR) and was calculated from the Investigator's assessment of response per RECIST 1.1 criteria. . The confirmed CR or PR was derived using the following rules: confirmed CR - at least two determinations of CR at least 4 weeks apart before disease progression; confirmed PR - at least two determinations of PR or better at least 4 weeks apart before progression.
Time Frame: From enrollment/randomization to the end of study, approximately 5.6 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 17 | 15 | 10
Percentage of participants | 35.3 [14.2 to 61.7] | 33.3 [11.8 to 61.6] | 30.0 [6.7 to 65.3]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of subjects with a complete response (CR), partial response (PR), or maintaining stable disease (SD) for at least 24 weeks while on study according to the investigator assessment of response per RECIST 1.1 criteria. CR and PR are confirmed responses derived using the following rules: Confirmed CR - at least 2 determinations of CR at least 4 weeks apart before disease progression. Confirmed PR - at least 2 determinations of PR or better at least 4 weeks apart before progression.
Time Frame: From enrollment/randomization the end of study, approximately 5.6 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 17 | 15 | 10
Percentage of participants | 35.3 [14.2 to 61.7] | 46.7 [21.3 to 73.4] | 30.0 [6.7 to 65.3]

7. Secondary Outcome: Association Between Biomarkers and PFS
Description: Describe if changes of biomarker expression at disease progression from baseline correlate with PFS.
Time Frame: From randomization to disease progression or death, up to approx. 5.6 years
Population: The number of patients with available biomarker data at both baseline and at progression is very small within each treatment arm (Arm A: n=7, Arm B: n=5, Arm C: n=5). This number of subjects is insufficient for an analysis to establish a relationship between the changes in biomarker at disease progression and progression free survival and would be statistically inappropriate to fit a model correlating changes in biomarkers with progression free survival with so few patients.
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 0 | 0 | 0

8. Post Hoc Outcome: All-Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 168 weeks for Lapatinib, (treatment duration ranged from 151 to 164 weeks), 164 weeks for Trastuzumab (treatment duration ranged from 0 to 160 weeks), 168 weeks for Aromatase Inhibitors (treatment duration ranged from 9 to 164 weeks).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approx. 5.6 years.
Time Frame: On-treatment deaths: up to approx. 168 weeks, Total deaths: up to approx. 5.6 years
Population: Clinical Database Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) - Arm B | Non-HER2- Enriched - Arm C
Number analyzed (Participants) | 17 | 15 | 10
Participants
  Total Deaths | 11 | 9 | 6
  On-treatment deaths | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 168 weeks for lapatinib, for a maximum duration of 164 weeks for trastuzumab and for a maximum duration of 168 weeks for aromatase inhibitors (anastrozole, letrozole and exemestane.)
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- TRAS+CHEM±AI (HER2-Enriched) • ArmB: Trastuzumab in HER2 Enriched: In subjects with HER2-overexpressing MBC with a molecular subtype of HER2 Enriched, Trastuzumab (loading dose of 8 mg/kg followed by the maintenance dose of 6 mg/kg IV q3weekly) along with chemotherapy of the investigator's choice or Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly along with chemotherapy of the investigators choice. Subjects randomized to this arm and hormone receptor positive received an aromatase inhibitor at the discretion of the investigator.
- Non-HER2-Enriched - Arm C: Lapatinib 1000mg + Trastuzumab in Non- HER2 Enriched: In subjects with HER2-overexpressing MBC with a molecular subtype of Non- HER2 Enriched (luminal A, luminal B or Basal type), Lapatinib 1000mg once daily orally along with Trastuzumab (loading dose of 8 milligram/ kilogram (mg/kg) followed by the maintenance dose of 6 mg/kg Intravenous (IV) Every 3 weeks (q3weekly)) or Lapatinib 1000 milligram (mg) once daily orally along with Weekly Trastuzumab (loading dose of 4 mg/kg) followed by maintenance dose of 2 mg/kg IV weekly. For subjects who were hormone receptor positive, an aromatase inhibitor of the investigator's choice was required.
Arm/Group | LAP+TRAS±AI (HER2-Enriched) - Arm A | TRAS+CHEM±AI (HER2-Enriched) • ArmB | Non-HER2-Enriched - Arm C
All-Cause Mortality (participants affected / at risk) | 3/17 | 1/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/15 | 2/10
Other Adverse Events (participants affected / at risk) | 15/17 | 14/15 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAP+TRAS±AI (HER2-Enriched) - Arm A (N=17) | TRAS+CHEM±AI (HER2-Enriched) • ArmB (N=15) | Non-HER2-Enriched - Arm C (N=10)
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LAP+TRAS±AI (HER2-Enriched) - Arm A (N=17) | TRAS+CHEM±AI (HER2-Enriched) • ArmB (N=15) | Non-HER2-Enriched - Arm C (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 1 | 6
Nausea (Gastrointestinal disorders) | 1 | 5 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4
Asthenia (General disorders) | 3 | 4 | 2
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 4 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 2
Blood sodium decreased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02213042/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT02213042/SAP_001.pdf